CLINICAL TRIAL: NCT01798121
Title: A Randomized, Double-blind, Equivalence Study of Tuberculin Purified Protein Derivative in Comparison With a Reference Standard Tuberculin Purified Protein Derivative (PPD-S2) for Detection of Tuberculosis in Subjects With a Confirmed Diagnosis of Tuberculosis.
Brief Title: Equivalence Study of Tuberculin Purified Protein Derivative in Comparison With a Reference Standard (PPD-S2)
Acronym: 02
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: JHP Pharmaceuticals LLC (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: JHP-Aplisol-02
Record Dates: First submitted 2013-01-31; First posted 2013-02-25 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Tuberculosis Identification.
Keywords: PPD; Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Tuberculin; Reference Standards

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aplisol (Experimental): To compare new PPD to reference standard material
  Interventions: Biological: To compare new PPD to reference standard material; Biological: Reference standard
- Reference standard (Placebo Comparator): Response of standard material
  Interventions: Biological: To compare new PPD to reference standard material

INTERVENTIONS:
Biological: To compare new PPD to reference standard material — Aplisol@ will be compared to reference standard material
  Other Names: Aplisol@
Biological: Reference standard — Response of reference standard material compared to Aplisol@.
  Other Names: Tuberculin PPD Standard.
  Arms: Aplisol

SUMMARY:
A study to determine bioequivalence of PPD material versus Reference Standard.

DETAILED DESCRIPTION:
This study is a multicenter, double-blind, active-controlled parallel-group study to determine the bioequivalence of newly produced PPD material versus PPD-S2 in the detection of male and female subjects with current or previously diagnosed intrathoracic Mtb infection, as documented by a positive culture for Mtb (preferred method), by their primary care or attending physician and/or by the subject's current or prior medical records (ie, sensitivity determination).

ELIGIBILITY:
Inclusion Criteria:

1. Males or nonpregnant females age 18 to 60 years
2. Documented PPD reactivity of 5 to 21 mm in the past, documented in a medical record. Self-reported PPD reactivity will be acc
3. Give written informed consent to participate
4. Generally healthy, as determined by medical history and targeted physical examination, if indicated
5. Possess 2 forearms that are free of burns, scars, eczema, or any physical deformity, which could impair injection of study prepar
6. Comprehension of the study requirements; expressed availability for the required study period, including readings at the nomina

Exclusion Criteria:

1. Prior PPD test within the past 30 days
2. Subject is of childbearing potential and unable to use contraceptives; is planning pregnancy; is pregnant or lactating
3. History of anaphylactic reaction, severe positive tuberculin reaction (eg, ulceration, necrosis) or other severe reaction to PPD in
4. Subject received a Bacillus Calmette-Guérin (BCG) vaccination in the past, or was born or lived outside the US as a child and is
5. Presence of conditions that may suppress TST reactivity -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-03 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Compare new PPD to Reference Standard | 72 hours
  Determine bio-equivalence of material used in trial by means of dose response and reaction sizes in patients.